CLINICAL TRIAL: NCT06530602
Title: Effect of 3-Dimensional Shoulder Complex Pain Alignment (3-D SPA) Mobilization on Frozen Shoulder.
Brief Title: 3-Dimensional Shoulder Complex Pain Alignment (3-D SPA) Mobilization on Frozen Shoulder.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Muniba
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Frozen Shoulder
Keywords: Frozen shoulder; QOL; Clinical trail; 3 D SPA; SPADI
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 3-D SPA (shoulder complex pain alignment) Moblization. Conventional therapy & Home Plan Treatment session: 3 per week, mobilization for 5 mins and 30 min session for total 3 weeks , exercises 3 sets for 10 repetitions.
  Modality: Ultrasound Mode: continuous 3 MHz, 1.5 w/cm2 for 6 min
  Interventions: Other: 3 D SPA (shoulder complex pain alignment) Moblization
- Group B (Active Comparator): Shoulder mobilization (kaltenborn) Conventional therapy & Home Plan Treatment session: 3 per week, mobilization for 5 mins and 30 min session for total 3 weeks , exercises 3 sets for 10 repetitions.
  Modality: Ultrasound Mode: continuous 3 MHz, 1.5 w/cm2 for 6 min
  Interventions: Other: Shoulder Moblization (KaltenBorn)

INTERVENTIONS:
Other: 3 D SPA (shoulder complex pain alignment) Moblization — 3 per week, mobilization for 5 mins and 30 min session for total 3 weeks , exercises 3 sets for 10 repetitions.
  Arms: Group A
Other: Shoulder Moblization (KaltenBorn) — 3 per week, mobilization for 5 mins and 30 min session for total 3 weeks , exercises 3 sets for 10 repetitions.
  Arms: Group B

SUMMARY:
Ongoing research aims to assess the enhancement of shoulder mobility by specifically addressing restrictions in all three planes of movement. current studies seek to investigate the impact of three-dimensional mobilization technique on their recovery and to prevent progression of disease to reduce pain, alleviate muscle tightness, facilitate tissue healing, and ultimately improve the range of motion in patients. A randomized control trial that will include total 36 participants. The first group will receive 3 Dimensional shoulder pain alignment (3-D SPA) mobilization along with conventional therapy and 2nd group will receive Shoulder mobilization along with conventional therapy. Data collected will be analyzed through SPSS 27.

DETAILED DESCRIPTION:
Decrease capacity of non contractile tissue ( such as joint capsule ) inflammation of capsule and ligament adhesion affects the shoulder joint, triggering stiffness and pain in Frozen shoulder. About 2% to 5% of the general population reported frozen shoulder without well known cause defined ,out of which Female patients 35 - 65 years of age.

hindrance in quality of life reported with performance of basic activities of daily living due to pain that worsen with movement and specifically at night , stiffness that cause mobility deficit.70% of female population are prone to get frozen shoulder. When reaching overhead, the arm is lifted by movements in the sternoclavicular , acromioclavicular (AC), scapulothoracic (ST), and gleno-humeral joints while overhead activities got limited in frozen shoulder.

Abnormal glenohumeral rhythm at scapulothoracic joint by posterior tilting of scapula and early upward motion of scapula occur. hence a capsular pattern developed in patient that comprise of External rotation, Abduction and Internal rotation.

Physiotherapy encompassed variety of treatment protocols for frozen shoulder including therapeutic modalities and manual therapy technique's consisting moblization, muscle energy techniques ,spencer's technique ,PNF and some of invasive treatments dry needling and therapeutic exercises.

3 D SPA is latest technique with no literature available for this to be applied to check its effectiveness on frozen shoulder rather it merely applied for post stroke shoulder pain prior in clinical setting . In group A 3-D SPA Moblization is employed that target moblization of AC joint (mobilizing it upward posteriorly) synchronously Scapula mobilized (abduction-adduction, anterior-posterior tilting) with glenohumeral Active motion in (flexion, horizontal abduction, horizontal adduction & External Internal rotation) all at once in all 3 planes frontal, sagittal, transverse plane while kaltenborn mobilization in anterior, posterior and inferior direction that is employed in group B, that has been a treatment of choice over the time is effective to treat frozen shoulder.

the study aim to evaluate the effect of 3-Dimensional Shoulder complex Pain Alignment (3-D SPA) mobilization technique on pain, disability, Range of Motion and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Local shoulder pain, often present either above the antero-medial and Lateral aspect of the shoulder.
* Stage II& III unilateral frozen shoulder Symptoms.
* Marked loss Of AROM & PROM with at least 50%loss of external rotation.
* Positive Apley's Scratch test.

Exclusion Criteria:

* Radiculopathy.
* Thoracic-outlet syndrome.
* Fractures and tumors of the upper extremity.
* Neurological disorders causing muscle weakness in the shoulder.
* Corticosteroid injection for frozen shoulder in last 3 months.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index | 3rd week
  Questionnaire comprise of 13 items evaluates both the degree of pain and the level of challenge in performing activities of daily living (ADLs) that involve the use of the upper extremities. The pain subscale comprises 5 items, while the Disability subscale consists of 8 items.
Measure Shoulder Range of Motion in Flexion | 3rd week
  changes from baseline ROM of shoulder flexion taken with goniometer
Measure Shoulder Range of Motion in Extension | 3rd week
  changes from baseline ROM of shoulder extension taken with goniometer
Measure Shoulder Range of Motion in abduction | 3rd week
  changes from baseline ROM of shoulder abduction taken with goniometer
Measure Shoulder Range of Motion in Horizontal abduction | 3rd week
  changes from baseline ROM of shoulder horizontal abduction taken with goniometer
Measure Shoulder Range of Motion in adduction | 3rd week
  changes from baseline ROM of shoulder adduction taken with goniometer
Measure Shoulder Range of Motion in horizontal adduction | 3rd week
  changes from baseline ROM of shoulder horizontal adduction taken with goniometer
Measure Shoulder Range of Motion in Internal rotation | 3rd week
  changes from baseline ROM of shoulder Internal rotation taken with goniometer
Measure Shoulder Range of Motion in External rotation | 3rd week
  changes from baseline ROM of shoulder External rotation taken with goniometer
Visual Analysis Scale | 3rd week
  Maximum score 10 minimum score 0 , it is used for both acute and chronic pain.

SECONDARY OUTCOMES:
WHOQoL-BREF | 3rd week
  Measures perception of life quality in four dimensions including physical, psychological, social relationship & environmental.
Apley's Scratch Test | 3rd week
  to check movements in all functional planes for the shoulder.

CONTACTS AND LOCATIONS:
Overall Officials: Madiha Ali, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No